CLINICAL TRIAL: NCT04224961
Title: Moderate Intensity Respiratory Muscle Training (RMT) in ALS
Brief Title: Respiratory Muscle Training (RMT) in ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00103777
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: ALS
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Minimal to No Respiratory Weakness (Experimental): MIP ≥ 70% predicted Complete home-based RMT program and participate in weekly web-based RMT therapy sessions.
  Interventions: Device: Respiratory Muscle Training
- Mild to Moderate Inspiratory Weakness (Experimental): MIP 40-70% predicted Complete home-based RMT program and participate in weekly web-based RMT therapy sessions.
  Interventions: Device: Respiratory Muscle Training

INTERVENTIONS:
Device: Respiratory Muscle Training — Two commercially available pressure-threshold RMT devices that utilize a spring-loaded flange to provide resistance against inspiration and expiration independent of respiratory flow rate will be used to provide the necessary range of resistance. Each participant will use two RMT devices, one for IMT and one for EMT.
  Other Names: EMST 150; Threshold IMT

SUMMARY:
Twelve adults with ALS will participate in a study involving four 3-week cycles of progressive respiratory muscle training (RMT). The investigators will measure maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) weekly. The investigators will obtain the majority of measurements of MIP and MEP during web-based telehealth visits. Participants will be stratified into 2 groups based on baseline inspiratory muscle strength as determined by maximum inspiratory pressure (MIP): six participants with minimal to no respiratory weakness (i.e., MIP ≥ 70% predicted) and six participants with mild to moderate inspiratory weakness (i.e., MIP 40-70% predicted).

DETAILED DESCRIPTION:
Twelve adults will participate in a single- subject A1-B-A2 study involving 4 visits to Duke over 24 weeks. The 6 week delayed start period (A1) will establish baseline status prior to initiation of RMT (B) and the follow-up period (A2) will determine detraining effects over 6 weeks of RMT withdrawal. Participants will complete four 3-week cycles of progressive RMT during the B phase. The investigators will measure MIP and MEP weekly. To reduce participant burden and enhance our ability to obtain repeated measures, the investigators will obtain 21 of 25 measurements of MIP and MEP during web-based telehealth visits.

Participants will complete a full assessment during the first study visit (M1) and receive training/instruction for obtaining MIP and MEP measurements at home with a portable, battery-powered digital pressure gauge manometer (MicroRPM Pressure Meter; Micro Direct). They will return to Duke for the pretest visit (M7), at which time a full assessment will be completed and RMT will commence. During the B phase, participants will complete 12-weeks of moderate intensity RMT, divided into four 3-week cycles, and participate in weekly web-based RMT therapy visits (M8-M18). Post-test assessment (M19) will occur immediately following completion of the 12-week RMT regimen. The investigators will measure MIP and MEP during RMT withdrawal via web-based telehealth visits (M20-24). Following the fourth and final on-site full assessment visit (M25), participants will return all equipment and will be offered the opportunity to initiate a clinical RMT regimen and receive follow-up care by Speech Pathology during future ALS Clinic visits.

Participants will be stratified into 2 groups based on baseline inspiratory muscle strength as determined by maximum inspiratory pressure (MIP): six participants with minimal to no respiratory weakness (i.e., MIP ≥ 70% predicted) and six participants with mild to moderate inspiratory weakness (i.e., MIP 40-70% predicted).

The primary outcomes are MIP and MEP. Secondary outcomes include peak cough flow (PCF) and sniff nasal inspiratory pressure (SNIP). Exploratory outcomes include the Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS), Eating Assessment Tool - 10 Item (EAT-10), 36-Item Short Form Survey (SF36), World Health Organization Quality of Life-BREF (WHOQOL-BREF), and Communicative Effectiveness Survey-Revised (CES-R). Clinical spirometry data will be extracted from the participant's electronic medical record if available from a coinciding ALS Clinic visit that occurs +/- 5 days from the assessment visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of ALS
* Ability to follow directions for study participation
* Ability to successfully and independently complete RMT repetitions at a minimum pressure-threshold target equal to 30% of MIP or MEP
* Ability to complete telehealth visits using a smartphone or computer with video capabilities
* Ability to complete a home-RMT regimen

Exclusion Criteria:

* MIP < 40 cmH20
* Presence of a tracheostomy
* Use of non-invasive or invasive ventilation when awake
* Participant or caregiver(s) inability to manipulate respiratory pressure meter, the RMT device, or calibration equipment for home training
* Inability to complete RMT repetitions successfully
* Concomitant neurologic or neurodegenerative conditions (e.g. stroke, dementia) or other serious conditions that would prevent meaningful study participation as determined at the discretion of the principal investigator
* Inability to give legally effective consent
* Inability to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Jones, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Minimal to No Respiratory Weakness: Maximum inspiratory pressure (MIP) ≥ 70% predicted. Complete home-based respiratory muscle training (RMT) program and participate in weekly web-based RMT therapy sessions.
  Respiratory Muscle Training: Two commercially available pressure-threshold RMT devices that utilize a spring-loaded flange to provide resistance against inspiration and expiration independent of respiratory flow rate will be used to provide the necessary range of resistance. Each participant will use two RMT devices, one for inspiratory muscle training (IMT) and one for expiratory muscle training (EMT).
- Mild to Moderate Inspiratory Weakness: MIP 40-70% predicted. Complete home-based RMT program and participate in weekly web-based RMT therapy sessions.
  Respiratory Muscle Training: Two commercially available pressure-threshold RMT devices that utilize a spring-loaded flange to provide resistance against inspiration and expiration independent of respiratory flow rate will be used to provide the necessary range of resistance. Each participant will use two RMT devices, one for IMT and one for EMT.
Period: Overall Study
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness
Started | 8 | 1
Completed | 7 | 0
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness | Total
Number analyzed (Participants) | 8 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.7) | 73.0 (0) | 62.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 1 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Safe, Well-tolerated Moderate Intensity Respiratory Muscle Training (RMT) as Measured by Rating of Perceived Exertion (RPE)
Description: Safe, well-tolerated moderate intensity Respiratory Muscle Training (RMT) is in part defined as an RPE between 4-5 and <6. The RPE is a way of measuring physical activity intensity level. Perceived exertion is how hard the participant feels like their body is working. 0 = rest, 1 = very easy, 2 = easy, 3 = moderate, 4 = somewhat hard, 5 = hard, 6 = harder, 7 = very hard, 8/9 = extremely hard, 10 = maximal.
Time Frame: 12 weeks
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness
Number analyzed (Participants) | 7 | 0
Participants | 4 |

2. Primary Outcome: Number of Participants With Safe, Well-tolerated Moderate Intensity Respiratory Muscle Training (RMT) as Measured by Pain Score
Description: Safe, well-tolerated moderate intensity Respiratory Muscle Training (RMT) is in part defined as a pain rating of <4 on a standard 0-10 scale, where 0 = no pain and 10 = the worst pain possible.
Time Frame: 12 weeks
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness
Number analyzed (Participants) | 7 | 0
Participants | 6 |

3. Primary Outcome: Number of Participants Able to Complete Respiratory Muscle Training (RMT)
Description: Feasibility will be determined by the number of participants able to complete the Respiratory Muscle Training
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness
Number analyzed (Participants) | 8 | 1
Participants | 7 | 0

4. Primary Outcome: Magnitude of Change in Maximum Inspiratory Pressure From Pre-test to Post-test as Determined by Cohen's Measure of Effect Size
Description: Magnitude of change for our primary outcome measures will be determined using Cohen's measure of effect size (d) as defined by the first equation for single-subject d provided by Busk and Serlin (1992). Simply stated, d is obtained by subtracting the mean of the first assessment from the mean of the second assessment, divided by the standard deviation of the first assessment. Effect size calculations will be determined to compare results from pre-test (M7) to post-test (M18). The investigators will use conservative interpretation guidelines for effect size calculations in which d < 0.6 is negligible, d ≥ 0.6 modest, d ≥ 1.0 large, and d ≥ 2.0 very large.
Time Frame: from pre-test (week 7) to post-test (week 18)
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness
Number analyzed (Participants) | 7 | 0
Participants
  Negligible | 5 |
  Modest | 1 |
  Large | 1 |

5. Primary Outcome: Magnitude of Change in Maximum Expiratory Pressure From Baseline to Withdrawal as Determined by Cohen's Measure of Effect Size
Description: Magnitude of change for our primary outcome measures will be determined using Cohen's measure of effect size (d) as defined by the first equation for single-subject d provided by Busk and Serlin (1992). Simply stated, d is obtained by subtracting the mean of the first assessment from the mean of the second assessment, divided by the standard deviation of the first assessment. Effect size calculations will be determined to compare results from baseline (M0-M5) to withdrawal (M19-M24). The investigators will use conservative interpretation guidelines for effect size calculations in which d < 0.6 is negligible, d ≥ 0.6 modest, d ≥ 1.0 large, and d ≥ 2.0 very large.
Time Frame: from baseline to withdrawal (up to week 24)
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness
Number analyzed (Participants) | 7 | 0
Participants
  Negligible | 5 |
  Large | 2 |

6. Secondary Outcome: Change in Peak Cough Flow in L/Min
Description: Effective peak cough flow in healthy subjects exceeds values of 360 to 400 L/min. PCF is measured at baseline, visit 7, visit 18 and visit 24. The overall change from baseline to visit 24 will be measured.
Time Frame: Baseline, 7 weeks, 18 weeks, 24 weeks
Population: Data not collected due to COVID restrictions, which prevented study staff from accessing the participants in order to perform the measurement. There are no plans to collect this data in the future.
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Sniff Nasal Inspiratory Pressure
Description: The sniff nasal inspiratory pressure (SNIP) consists in the measurement of pressure through an occluded nostril during sniffs performed through the contralateral nostril. SNIP is measured through a plug occluding one nostril during sniffs through the contralateral nostril. A plateau in pressure is reached after 5-10 sniffs in most individuals 1. For SNIP measurement, 10 sniffs are usually performed. The SNIP is measured at baseline, visit 7, visit 18 and visit 24. The overall change from baseline to visit 24 will be measured.
Time Frame: Baseline, 7 weeks, 18 weeks, 24 weeks
Population: as for outcome 6
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to approximately 24 weeks
Description: Adverse events/serious adverse events were systematically investigated at each study visit and recorded using REDCap.
Arm/Group | Minimal to No Respiratory Weakness | Mild to Moderate Inspiratory Weakness
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/1
Other Adverse Events (participants affected / at risk) | 5/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minimal to No Respiratory Weakness (N=8) | Mild to Moderate Inspiratory Weakness (N=1)
Respiratory decline (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minimal to No Respiratory Weakness (N=8) | Mild to Moderate Inspiratory Weakness (N=1)
Dysphonia (General disorders) | 0 | 1
Neck weakness/tightness (Musculoskeletal and connective tissue disorders) | 1 | 1
Seasonal allergies/headache (General disorders) | 1 | 0
Dizziness (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
COVID diagnosis (Infections and infestations) | 1 | 0
Fall without injury (General disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT04224961/Prot_SAP_000.pdf